CLINICAL TRIAL: NCT02252679
Title: Endogenous Calcium Stable Isotope Study (eCaSIS): Evaluation of MC-ICP-MS as a Diagnostic Tool for Metabolic Bone Diseases and Disorders of Calcium Metabolism
Brief Title: Study of the Diagnostic Value of Stable Calcium Isotope Profiling in Bone and Calcium Disorders
Acronym: eCaSIS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: GEOMAR-Helmholtz Centre for Ocean Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: UZ Leuven - s56719
Record Dates: First submitted 2014-09-22; First posted 2014-09-30 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Bone Diseases; Osteomalacia; Osteoporosis
Keywords: Bone Turnover Markers; Calcium Isotopes
MeSH Terms: conditions — Bone Diseases; Osteomalacia; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, spot urine and/or 24h urine collection samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Osteoporosis: Postmenopausal women, men > age 50 years, or other patients with well-established causes of secondary osteoporosis (incl. glucocorticoid-induced osteoporosis, transplantation-related osteoporosis, disuse osteoporosis, etc.) N=20 treated with antiresorptive drugs N=10 treated with osteoanabolic drugs (e.g. teriparatide, Forsteo)
- Calcium malabsorption: N=10 Patients with clinically obvious potential causes of calcium malabsorption (incl. severe vitamin D-deficiency, Scopinaro or other bariatric surgery, exocrine pancreatic insufficiency/steatorrhea, cystic fibrosis, inflammatory bowel disease, celiac disease, anorexia nervosa/eating disorders, malnutrition, etc.), with or without bone pains, muscle weakness and other typical osteomalacia symptoms. Confirmed by 24h urine collection showing calciuria <100 mg/24h.
- Various disorders: Exploratory, heterogeneous group of calcium-related disorders (incl.hypercalcemia, hypocalcemia, primary/secondary/tertiary hyperparathyroidism, hypoparathyroidism, vitamin D deficiency, X-linked/autosomal dominant hypophosphatemic rickets, familial hypocalciuric hypocalcemia,etc.) N=20
- Normal control subjects: N=40 Men and women ≤ 40 years recruited from the population

SUMMARY:
The purpose of this study is to determine whether mass spectrometry analysis of stable (non-radioactive) calcium isotopes in plasma or urine samples can help in the diagnosis of bone and calcium disorders.

DETAILED DESCRIPTION:
The aim of this pilot study is to explore the diagnostic value of MC-ICP-MS (multicollector inductively coupled plasma mass spectrometry) or TIMS (thermal ionization mass spectrometry) measurement of endogenous stable calcium isotopes in plasma and urine samples in patients seen during routine clinical care at the outpatient clinics (incl. Center for Metabolic Bone Diseases) of the University Hospitals Leuven.

ELIGIBILITY:
Inclusion Criteria:

* DXA (dual energy X-ray absorptiometry) T-score known clinically to be = or < -2.5 OR presence of low-energy osteoporotic fractures (i.e. excluding those of the skull, fingers and toes) [for osteoporosis and calcium malabsorption patients]

Exclusion Criteria:

* inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinical convenience sample Healthy volunteers recruited from the communities in Leuven and neighbouring cities Siblings, parents or other relatives of patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Likelihood ratio (LR) of urinary calcium δ44/40 Ca (‰) values for diagnosing negative skeletal calcium balance | follow-up will vary on clinical basis, with expected averages of 1 year (for osteoporosis) to 3 months (for other conditions)
  The sensitivity, specificity, positive and negative predictive value of the new test will be compared to expert clinical diagnosis as the gold standard. This diagnosis is established during follow-up and based on clinical observations, bone mineral density results/changes, bone turnover markers and response to treatments.

SECONDARY OUTCOMES:
Likelihood ratio (LR) of plasma calcium δ44/40 Ca (‰) values for diagnosing negative skeletal calcium balance | follow-up will vary on clinical basis, with expected averages of 1 year (for osteoporosis) to 3 months (for other conditions)
  The sensitivity, specificity, positive and negative predictive value of the new test will be compared to expert clinical diagnosis as the gold standard. This diagnosis is established during follow-up and based on clinical observations, BMD results, bone turnover markers and response to treatments.
Area under the receiver-operator curve (AUROC) of calcium δ44/40 Ca (‰) values compared to bone turnover markers, with expert clinical diagnosis as the golden standard | follow-up will vary on clinical basis, with expected averages of 1 year (for osteoporosis) to 3 months (for other conditions)
  Osteocalcin and bèta-CTx (C-terminal telopeptide of type I collagen) will be measured.

OTHER OUTCOMES:
Inter- and intra-assay variability of plasma and urine calcium δ44/40 Ca (‰) values | follow-up will vary on clinical basis, with expected averages of 1 year (for osteoporosis) to 3 months (for other conditions)
calcium δ44/40 Ca (‰) values of human bone samples | before and 1 year after kidney transplantation
  Secondary use of bone biopsy samples obtained in the Leuven Bone Biopsy Program (NCT01886950)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Vanderschueren, MD, PhD, Principal Investigator — UZ Leuven
Locations (2):
- UZ Leuven, Leuven, Belgium
- GEOMAR-Helmholtz Centre for Ocean Research, Kiel, Germany

REFERENCES:
- [Background] Khalil R, Antonio L, Laurent MR, David K, Kim NR, Evenepoel P, Eisenhauer A, Heuser A, Cavalier E, Khosla S, Claessens F, Vanderschueren D, Decallonne B. Early effects of androgen deprivation on bone and mineral homeostasis in adult men: a prospective cohort study. Eur J Endocrinol. 2020 Aug;183(2):181-189. doi: 10.1530/EJE-20-0348. PMID 32454455